CLINICAL TRIAL: NCT03695835
Title: A Retrospective and Prospective Study of a New Immunotherapy Regimen (MyVaccx) for Patients With Adenocarcinoma.
Brief Title: A Data Collection Study for Patients With Adenocarcinoma Treated With the MyVaccx Immunotherapy Regimen.
Acronym: NIRPA
Status: Completed | Type: Observational
Sponsor: Gary Onik MD (Individual)
Responsible Party: Sponsor
Other Study IDs: NIRPA
Record Dates: First submitted 2018-09-28; First posted 2018-10-04 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Adenocarcinoma
Keywords: prostate cancer; lung cancer; pancreatic cancer; colorectal cancer; bladder cancer
MeSH Terms: conditions — Adenocarcinoma; Prostatic Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Urinary Bladder Neoplasms | interventions — Ipilimumab; pembrolizumab; sargramostim

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adenocarcinoma treated with MyVaccx: MyVaccx combines tumor ablation and immunotherapeutic agents for treatment of late stage cancer disease..
  Interventions: Drug: Immunotherapeutic Agents; Device: Ablation

INTERVENTIONS:
Drug: Immunotherapeutic Agents — Antigen exposure immediately followed by in situ injection of combination of immunotherapeutic agents
  Other Names: Yervoy, Keytruda, Leukine
Device: Ablation — Antigen exposure immediately followed by in situ injection of combination of immunotherapeutic agents
  Other Names: Cryo and radio frequency (RF) ablation

SUMMARY:
A retrospective and prospective data collection study on 27 consecutive subjects with adenocarcinoma who were treated using the MyVaccx system by Dr. Gary Onik. Retrospective data were collected on the treatment with the immunotherapy system and prospective data will be collected as they are prospectively monitored through their normal standard of care for their original cancer.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with the MyVaccx System
* Greater than 18 years of age
* Signature of the informed consent

Exclusion Criteria:

* 2 subjects treated with the MyVaccx System with known visceral disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with adenocarcinoma treated with the MyVaccx System through the Center for High Risk and Recurrent Prostate Cancer.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
MyVaccx immunotherapy treatment impact on late stage cancer disease | From date of treatment until the date of death from any cause up to 60 months
  Time to death after the start of treatment

SECONDARY OUTCOMES:
MyVaccx immunotherapy treatment impact on late stage cancer disease | Time to progression after a complete or partial response up to 60 months
  Complete and partial response to treatment based on the iRESIST criteria

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for High Risk and Recurrent Prostate Cancer, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a medical journal.
Supporting Information: Study Protocol
Time Frame: After retrospective data collection is completed.

DOCUMENTS (1):
  • Study Protocol (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT03695835/Prot_000.pdf